CLINICAL TRIAL: NCT01746277
Title: A Phase Ⅱ Randomized Controlled Trial to Compare Chemotherapy Sequenced by EGFR-TKIs and Chemotherapy Combined With EGFR-TKIs for Advanced or Metastatic NSCLC Patients Failed to EGFR-TKIs Therapy
Brief Title: Study of Chemotherapy Sequenced by or Combined With EGFR-TKIs for NSCLC Patients Failed to EGFR-TKIs Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH S-462
Record Dates: First submitted 2012-12-04; First posted 2012-12-10 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: non small cell lung cancer; chemotherapy; epidermal growth factor receptor tyrosine kinase inhibitor; retreatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Pemetrexed; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- combined group (Other): combined group chemotherapy with docetaxel 75mg/m2 d1 or pemetrexed 500mg/m2 d1, every 3 weeks,at least 2 cycles and the maximal cycle is 6 depending on disease evaluation and patient's physical condition combined with gefitinib 250mg once per day from the start day of chemotherapy until disease progression or intolerable side effects.
  Interventions: Drug: combined group
- sequenced group (Other): sequenced group chemotherapy with docetaxel 75mg/m2 d1 or pemetrexed 500mg/m2 d1, every 3 weeks,at least 2 cycles and the maximal cycles is 6 depending on disease evaluation or patient's physical condition sequenced by gefitinib 250mg once per day until disease progression or intolerable side effects.
  Interventions: Drug: Sequenced group

INTERVENTIONS:
Drug: combined group — chemotherapy with docetaxel 75mg/m2 d1 or pemetrexed 500mg/m2 d1, every 3 weeks,at least 2 cycles and the maximal cycle is 6 depending on disease evaluation and patient's physical condition combined with gefitinib 250mg once per day from the start day of chemotherapy until disease progression or intolerable side effects.
  Other Names: Docetaxel (Taxotere); Pemetrexed (Alimta); Gefitinib (Iressa)
  Arms: combined group
Drug: Sequenced group — sequenced group chemotherapy with docetaxel 75mg/m2 d1 or pemetrexed 500mg/m2 d1, every 3 weeks,at least 2 cycles and the maximal cycles is 6 depending on disease evaluation or patient's physical condition sequenced by gefitinib 250mg once per day until disease progression or intolerable side effects.
  Other Names: Docetaxel (Taxotere); Pemetrexed (Alimta); Gefitinib (Iressa)
  Arms: sequenced group

SUMMARY:
There are two different treatment modes for NSCLC patients who failed to epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI) after initially responding to EGFR-TKI. One is EGFR-TKI combined with chemotherapy and the other is chemotherapy followed by EGFR-TKI. It is unclear which one is more suitable to this group of lung cancer patients. So this phase Ⅱclinical trial is designed to compare the efficiency and safety of these two different treatment modes.

DETAILED DESCRIPTION:
Responses to EGFR-TKIs are quiet dramatic and durable, especially in patients with EGFR gene classic mutations, such as 19 deletion or 21 leucine 858 arginine(L858R). However, most patients with NSCLC who respond to EGFR-TKIs eventually experience progression of disease after approximately 12 months. The lack of an established therapeutic option for NSCLC patients who have progressive disease after EGFR-TKIs failure poses a great challenge to physicians in terms of how best to manage this growing group of lung cancer patients.

In clinical practice some of the initially EGFR-TKI sensitive tumors which progressed evidence a striking increase in tumor volume within several weeks, after being taken off EGFR-TKI. This response is called "rebound phenomenon". Most experts still believe that these tumors continue to be "oncogene-addicted" to EGFR. So it is rational that EGFR-TKI combined with another chemotherapy regimen can be used to treat NSCLC after the failure of EGFR-TKI therapy.

However in some phase Ⅱclinical trials involved a few NSCLC patients who failed to EGFR-TKI therapy, another treatment mode, that is to say, at least one cytotoxic chemotherapy was used firstly then switched to EGFR-TKI therapy until progression of disease, was used and called reintroduction or retreatment of EGFR-TKI. Using this treatment mode, some investigators reported the partial remission (PR) and disease control rate (DCR) were observed in 21.7%-36% and 65.2%-86% NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* histologically and cytologically proven non-small cell bronchogenic carcinoma (sputum cytology alone was not acceptable)
* clinical stages ⅢB or Ⅳ
* recurrent or refractory disease following previous first-line chemotherapy regimens containing platinum and second-line EGFR-TKIs therapy
* partial remission (PR) or stable disease (SD) at least for 6 months during previous EGFR-TKI treatment
* at least one bidimensionally measurable or radiographically assessable lesion
* Eastern cooperative oncology group performance status (ECOG PS) ≤ 2
* life expectancy ≥ 12 weeks
* adequate hematological, renal, and hepatic functions

Exclusion Criteria:

* additional malignancies
* uncontrolled systemic disease
* any evidence of clinically active interstitial lung disease
* newly diagnosed central nervous system (CNS) metastasis and not treated by radiotherapy or surgery
* pregnancy or breast feeding phase

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-10 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
progression free survival | up to 52 weeks (about one year)
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 52 weeks.

SECONDARY OUTCOMES:
overall survival | up to 100 weeks
  From date of randomization until the date of death from any cause, assessed up to 100 weeks.
objective response rate | up to 9 weeks
  The objective response rate includes the complete remission and partial remission rate.
the score of functional assessment of cancer treatment-lung(FACT-L) | up to 100weeks
  FACL-L is assessed at different time points.(Date of randomization,1 week after chemotherapy,every cycle of chemotherapy,every month of EGFR-TKI maintain treatment,up to 100 weeks)
Number of participants with adverse events | Participants will be followed for the duration of treatment, an expected average of 52 weeks.
  The adverse events are assessed by National Cancer Institute-Common Toxicity Criteria(version3.0) (NCI-CTC).

CONTACTS AND LOCATIONS:
Overall Officials: Mengzhao Wang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Department of Respiratory Medicne, Peking Union Medical Hospital, Beijing, China

REFERENCES:
- [Result] Oh IJ, Ban HJ, Kim KS, Kim YC. Retreatment of gefitinib in patients with non-small-cell lung cancer who previously controlled to gefitinib: a single-arm, open-label, phase II study. Lung Cancer. 2012 Jul;77(1):121-7. doi: 10.1016/j.lungcan.2012.01.012. Epub 2012 Feb 12. PMID 22333554
- [Result] Li J, Hao X, Wang Y, Zhang X, Shi Y. [Clinical response to gefitinib retreatment of lung adenocarcinoma patients who benefited from an initial gefitinib therapy: a retrospective analysis]. Zhongguo Fei Ai Za Zhi. 2012 Jan;15(1):44-8. doi: 10.3779/j.issn.1009-3419.2012.01.09. Chinese. PMID 22237124
- [Result] Watanabe S, Tanaka J, Ota T, Kondo R, Tanaka H, Kagamu H, Ichikawa K, Koshio J, Baba J, Miyabayashi T, Narita I, Yoshizawa H. Clinical responses to EGFR-tyrosine kinase inhibitor retreatment in non-small cell lung cancer patients who benefited from prior effective gefitinib therapy: a retrospective analysis. BMC Cancer. 2011 Jan 1;11:1. doi: 10.1186/1471-2407-11-1. PMID 21194487
- [Result] Becker A, Crombag L, Heideman DA, Thunnissen FB, van Wijk AW, Postmus PE, Smit EF. Retreatment with erlotinib: Regain of TKI sensitivity following a drug holiday for patients with NSCLC who initially responded to EGFR-TKI treatment. Eur J Cancer. 2011 Nov;47(17):2603-6. doi: 10.1016/j.ejca.2011.06.046. Epub 2011 Jul 23. PMID 21784628